CLINICAL TRIAL: NCT02534584
Title: Impact of Compliance With a Care Bundle on Acute Kidney Injury Outcomes
Brief Title: Use of Care Bundle in Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr. Nitin Kolhe, Consultant Nephrologist, University Hospitals of Derby and Burton NHS Foundation Trust
Other Study IDs: 1.0
Record Dates: First submitted 2015-08-23; First posted 2015-08-27 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; outcome; mortality; care-bundle
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a service evaluation to assess the impact of compliance of Acute Kidney Injury care bundle (AKI-CB) on clinical and renal outcomes. The AKI care bundle is coupled with an interruptive electronic alert, which is triggered by the first attempt to order blood tests or medications on patients who have been identified as having AKI by the electronic recognition from serum creatinine results. The interruptive alert will warn the clinician about AKI and request them to complete the AKI care bundle. Once the AKI care bundle is completed, the clinician is able to request blood tests or medication. The clinician will be able to override the alert only after stating the reason. Education with respect to importance of AKI and the AKI-CB is provided every four months when junior doctors rotated through different specialities and also at clinical governance days. The investigators will compare AKI episodes, which have the AKI-CB completed early (defined as within 24 hours of availability of the blood results) with those who either had the AKI-CB completed late (defined as after 24 hours of availability of the blood results) or not completed at all. The AKI patients who either had the AKI-CB completed late or not completed will be considered as not having the AKI-CB completed for this analysis.

DETAILED DESCRIPTION:
This single centre study will be conducted at the Royal Derby Hospital, a 1139-bed tertiary care centre. Data will be collected from February 2013 to December 2013 on all adult patients over the age of 18 years. An electronic recognition system for AKI has been in use since 2010 that allows prospective data collection for all cases of AKI. The electronic recognition system was modified in December 2012, to incorporate the Kidney Diseases Improving Global Outcomes (KDIGO) definitions for AKI. In an effort to improve the clinical outcomes, intranet guidelines were introduced along with the electronic recognition and alerting system. In December 2012, a one-page paper version of the AKI CB was devised, which was subsequently incorporated into the hospital electronic patient record on 1st February 2013. During this period, education on the AKI CB was given to all staff in acute areas of the hospital and a poster explaining the AKI CB was displayed in all clinical areas. The hospital already has electronic ordering of investigations and prescribing of medications in place. The CB consists of simple standardized investigations and interventions, reminding clinicians of the importance of thorough Assessment, Urinalysis, establishing a Diagnosis, planning Investigations and Treatment and at the same time issuing guidance about Seeking advice from nephrologist while caring for patients with AKI (AUDITS). All the steps in the CB are objective and the clinicians are requested to click yes or no for each step of the CB. On 1st August 2013, the AKI CB was coupled with an interruptive electronic alert, which was triggered by the first attempt to order blood tests or medications on patients who had been identified as having AKI. The interruptive alert would warn the clinician about AKI and request them to complete the AKI CB. Once the AKI CB was completed, the clinician was able to request blood tests or medication. The clinician would be able to override the alert only after stating the reason. The location of patients was categorized into the following divisions - Medical Assessment Unit, Medical wards, Surgical & Orthopedic wards, Haematology and Oncology wards, Intensive Care and Surgical Step Down (high dependency unit) and Other wards.

A weekly report is automatically generated which captures patient location in the hospital, age, date of admission, date of discharge, finished consultant episode and survival status at the reporting date.

For this study, the investigators will analyze all AKI episodes, which had the AKI CB completed early (defined as within 24 hours of availability of the blood results) with those who either had AKI CB completed late (defined as after 24 hours of availability of the blood results) or not completed at all. The AKI episodes who either had AKI CB completed late or not completed will be considered as not having AKI CB completed for this analysis. Community acquired AKI will be defined as AKI within 24 hours of admission. Survival status of all patients will be obtained in February 2015.

ELIGIBILITY:
Inclusion Criteria:

* All episodes of acute kidney injury in adults patients

Exclusion Criteria:

* Age less than 17 years
* Patients without acute kidney injury

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adults patients with acute kidney injury
Sampling Method: Probability Sample
Enrollment: 944 (Actual)
Dates: Start 2013-08; Primary Completion 2015-01 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Mortality | 1 year
  This is the average follow up

SECONDARY OUTCOMES:
Length of stay | 10 days
  This is average length of stay
Severity of AKI as measured by AKI stages | 10 days
  Proportion of patients whose AKI increases in severity, from AKI stage 1 to stage 2 and from stage 2 to stage 3

CONTACTS AND LOCATIONS:
Overall Officials: Nitin V Kolhe, MD, DM, Principal Investigator — Derby Teaching Hospital NHS Trust
Locations (1):
- Derby Hospital NHS Foundation Trust, Derby, Derbyshire, United Kingdom